CLINICAL TRIAL: NCT07154745
Title: A Single Arm Study to Evaluate the Efficacy and Safety of Pozelimab and Cemdisiran Combination Therapy in Patients With Paroxysmal Nocturnal Hemoglobinuria With Inadequate Control of Intravascular Hemolysis on Currently Available C5 Inhibitor Therapy
Brief Title: A Study to Evaluate How Pozelimab + Cemdisiran Combination Therapy Works in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH) Whose Current Treatment is Not Working Efficiently
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R3918-PNH-2483; 2024-519709-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-13; First posted 2025-09-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pozelimab + Cemdisiran Combo (Experimental)
  Interventions: Drug: Pozelimab; Drug: Cemdisiran

INTERVENTIONS:
Drug: Pozelimab — Administered per the protocol
  Other Names: REGN3918
Drug: Cemdisiran — Administered per the protocol
  Other Names: ALN-CC5

SUMMARY:
This study is researching a treatment combination with two experimental drugs called pozelimab and cemdisiran referred to as "study drugs". Researchers are looking for a better way to treat Paroxysmal Nocturnal Hemoglobinuria (PNH).

The aim of the study is to see how well the pozelimab and cemdisiran combination works to lower hemolysis in participants whose PNH has been not well controlled even after taking other complement component 5 (C5) inhibitors, eculizumab/eculizumab biosimilar, ravulizumab or crovalimab.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drugs?
* How much of the study drugs are in the blood at different times?
* Whether the body makes antibodies against the study drug (which could make the study drugs not work as well or could lead to side effects)

DETAILED DESCRIPTION:
The treatment period has two parts, a Treatment Period (TP, 28 weeks) and an Extension treatment Period (EP, 52 weeks).

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of PNH confirmed by a history of high-sensitivity flow cytometry from prior testing
2. Currently treated with marketed eculizumab, ravulizumab, or crovalimab at the labeled dose for at least 6 months
3. LDH persistently > 1.5 × Upper Limit of Normal (ULN) in the previous 6 months that the Principal Investigator (PI) attributes is due to intravascular hemolysis
4. At least 2 screening LDH values from different visits as described in the protocol
5. Willing and able to comply with clinic/remote visits and study-related procedures, including completion of the full series of meningococcal vaccinations required per protocol and agreement to continue to remain up to date with these vaccinations during the study

Key Exclusion Criteria:

1. Receipt of an organ transplant, history of bone marrow transplantation or other hematologic transplants
2. Body weight <40 kilograms at screening visit
3. Patients with a known or suspected C5 mutation that is refractory to their current C5i treatment as described in the protocol
4. Any active or ongoing infection within 2 weeks of screening or during the screening period or any recent infection as described in the protocol
5. Known hereditary complement deficiency

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-09-08 (Estimated); Study Completion 2031-07-25 (Estimated)

PRIMARY OUTCOMES:
Percent change in Lactate Dehydrogenase (LDH) during TP | From baseline to week 28

SECONDARY OUTCOMES:
Normalization of LDH | Through week 52
Adequate control of hemolysis (LDH ≤1.5 × ULN) | Through week 52
Transfusion avoidance | Through week 52
  Not requiring a Red Blood Cell (RBC) transfusion as per protocol algorithm based on hemoglobin values
Hemoglobin stabilization | Through week 52
  Participants who do not receive an RBC transfusion and have no decrease in hemoglobin level of ≥2 g/dL
Change in hemoglobin from baseline | Through week 52
Change in fatigue | Through week 52
  As measured by the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale.
  The FACIT-Fatigue assesses the level of fatigue using a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). Scores range from 0 to 52, with higher scores indicating a higher quality of life
Occurrence of all Adverse Events (AEs) | Through week 52
Severity of all AEs | Through week 52
Occurrence of all Treatment-Emergent Adverse Events (TEAEs) | Through week 52
Severity of all TEAEs | Through week 52
Change from baseline in Total Complement Hemolytic Activity Assay (CH50) | Through week 52
Concentrations of total pozelimab | Through week 52
Concentrations of cemdisiran | Through week 52
Concentrations of total C5 | Through week 52
Incidence of Anti-Drug Antibody (ADA) to pozelimab | Through week 52
Magnitude of ADA to pozelimab | Through week 52
Incidence of ADA to cemdisiran | Through week 52
Magnitude of ADA to cemdisiran | Through week 52
Percent change in LDH during EP | From baseline to week 24 and week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/